CLINICAL TRIAL: NCT01554241
Title: Optimizing Vitamin D in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DinNH2012; 1R21AG04166001-A1 (Other Grant/Funding Number: National Institute on Aging); additional funder (Other Grant/Funding Number: 1R21AG04166001-A1 Office of Dietary Supplements)
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Deficiency of Vitamin D3
Keywords: vitamin D3; D3; cholecalciferol; 25-OH vitamin D; elderly; nursing home resident
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- vitamin D3 800 IU/day (Experimental): recommended daily dosage of 800 IU/day D3
  Interventions: Dietary Supplement: vitamin D3 800 IU/day
- 2000 IU/day D3 (Experimental): D3 2000 IU/day
  Interventions: Dietary Supplement: D3 2000 IU/day
- vitamin D3 4000 IU/day (Experimental): D3 4000 IU/day
  Interventions: Dietary Supplement: D3 4000 IU/day
- 50,000 IU/week D3 (Experimental): D3 50,000 IU weekly
  Interventions: Dietary Supplement: D3 50,000 IU weekly

INTERVENTIONS:
Dietary Supplement: D3 2000 IU/day — 2000 IU/day D3
  Other Names: cholecalciferol
  Arms: 2000 IU/day D3
Dietary Supplement: D3 4000 IU/day — vitamin D3 4000 IU/day
  Other Names: cholecalciferol
  Arms: vitamin D3 4000 IU/day
Dietary Supplement: D3 50,000 IU weekly — vitamin D3 50,000 IU/week
  Other Names: cholecalciferol
  Arms: 50,000 IU/week D3
Dietary Supplement: vitamin D3 800 IU/day — vitamin D3 800 IU/day
  Other Names: cholecalciferol
  Arms: vitamin D3 800 IU/day

SUMMARY:
Vitamin D deficiency is highly prevalent in older people in the absence of vitamin D supplementation. The limited data available show marked inter-individual variability in response to vitamin D supplementation in very old, frail elderly with almost 25% remaining vitamin D deficient (25-OH D < 20 ng/mL) when receiving the currently recommended 800 IU/day vitamin D. This proposal is for exploratory research on the use of a wide range of oral vitamin D3 doses in frail elderly living in controlled living environments.

DETAILED DESCRIPTION:
The investigators will determine the dose response relationship of circulating total and unbound 25-OH vitamin D3 to supplemental vitamin D3 at daily doses of 800 (currently recommended for the elderly), 2000, and 4000 IU or 50,000 IU/weekly in a randomized blinded investigation of 16 weeks duration. The investigators will also compare the efficacy of each dosing regimen in achieving 25-OH vitamin D levels >20 ng/mL (50 nmol/L) and identify covariates that contribute to inter-individual variation in the dose response relationship. In patients with osteoporosis, relationships between unbound vs. total 25-OH on intact parathyroid hormone and a marker of bone resorption (beta-Ctx) will be analyzed. The investigators will also examine responses of inflammatory cytokines.

Note: as of April 8,2014, there will be no further enrollment in the 50,000 IU/weekly dose group

ELIGIBILITY:
Inclusion Criteria:

* age over 65
* medically stable
* residing in long-term care or assisted living

Exclusion Criteria:

* hypercalcemia or high risk for hypercalcemia
* active cancer or malignancy other than non-melanoma skin cancer
* severe renal disease (eGFR <30 ml/mkin/M2)
* small bowel resection or intestinal bypass surgery
* hyperparathyroidism
* granulomatous disease
* clinically unstable (changes in medications or diagnoses within a month, hospitalizations, within 6 months)
* allergy to vitamin D

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice B Schwartz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following participant consent/enrollment, 4 were ineligible due to clinical instability or abnormal laboratory tests and one withdrew consent.
Period: Overall Study
Arm/Group | Vitamin D3 800 IU/Day | 2000 IU/Day D3 | Vitamin D3 4000 IU/Day | 50,000 IU/Week D3
Started | 23 | 20 | 24 | 14
Completed | 20 | 19 | 20 | 13
Not Completed | 3 | 1 | 4 | 1
Not completed — Death | 3 | 1 | 1 | 0
Not completed — protocol specified renal stone | 0 | 0 | 0 | 1
Not completed — protocol specified change in eGFR | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Elderly (>65 yr) clinically stable long-term stay nursing home residents with no contraindications or allergy to D, osteoporosis or a history of fractures and receiving over 800 IU/day D, treatment for severe D deficiency or investigational agent in the prior six months on no D or had stable D doses for over two months .
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 800 IU/Day | 2000 IU/Day D3 | Vitamin D3 4000 IU/Day | 50,000 IU/Week D3 | Total
Number analyzed (Participants) | 23 | 20 | 24 | 14 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 23 | 20 | 24 | 14 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.9 (8.7) | 85.9 (8.5) | 89.5 (6.6) | 90.1 (6.6) | 87.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 16 | 10 | 52
  Male | 10 | 7 | 8 | 4 | 29
Region of Enrollment [Number; unit: participants]
  United States | 23 | 20 | 24 | 14 | 81

OUTCOME MEASURES:

1. Primary Outcome: Total 25-OH Vitamin D3 Level
Description: circulating total 25-OH vitamin D concentration
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D3 800 IU/Day | 2000 IU/Day D3 | Vitamin D3 4000 IU/Day | 50,000 IU/Week D3
Number analyzed (Participants) | 20 | 19 | 20 | 13
ng/mL | 33 (6) | 34 (6) | 43 (10) | 61 (14)
Statistical Analysis 1: Comparison: Vitamin D3 800 IU/Day vs 2000 IU/Day D3 vs Vitamin D3 4000 IU/Day vs 50,000 IU/Week D3; Comparisons of concentrations in D3 dosing groups at study end were made by ANOVA. Adherence of 80% was pre-specified for inclusion in analyses; Test type: Superiority or Other; p < .0001, ANOVA; Results presented were Bonferonni-corrected for a mid-point safety analysis
Statistical Analysis 2: Comparison: Vitamin D3 800 IU/Day vs 2000 IU/Day D3; Test type: Superiority or Other; p = .56, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 3: Comparison: Vitamin D3 800 IU/Day vs Vitamin D3 4000 IU/Day; Test type: Superiority or Other; p < .0009, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 4: Comparison: Vitamin D3 800 IU/Day vs 50,000 IU/Week D3; Test type: Superiority or Other; p < .0001, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 5: Comparison: 2000 IU/Day D3 vs Vitamin D3 4000 IU/Day; Test type: Superiority or Other; p < .006, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 6: Comparison: 2000 IU/Day D3 vs 50,000 IU/Week D3; Test type: Superiority or Other; p < .0001, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 7: Comparison: Vitamin D3 4000 IU/Day vs 50,000 IU/Week D3; Test type: Superiority or Other; p < .0001, ANOVA; Bonferroni/Dunn adjustment

2. Secondary Outcome: Free 25-OH Vitamin D3
Description: circulating free 25-OH vitamin D3 concentration
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vitamin D3 800 IU/Day | 2000 IU/Day D3 | Vitamin D3 4000 IU/Day | 50,000 IU/Week D3
Number analyzed (Participants) | 20 | 19 | 20 | 13
pg/mL | 8.7 (2.1) | 9.5 (1.7) | 12.2 (4.3) | 16.8 (4.3)
Statistical Analysis 1: Comparison: Vitamin D3 800 IU/Day vs 2000 IU/Day D3 vs Vitamin D3 4000 IU/Day vs 50,000 IU/Week D3; Test type: Superiority or Other; p < .0001, ANOVA — analyses were corrected for multiple comparisons (Bonferroni)
Statistical Analysis 2: Comparison: Vitamin D3 800 IU/Day vs 2000 IU/Day D3; Test type: Superiority or Other; p = 0.47, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 3: Comparison: Vitamin D3 800 IU/Day vs Vitamin D3 4000 IU/Day; Test type: Superiority or Other; p < .002, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 4: Comparison: Vitamin D3 800 IU/Day vs 50,000 IU/Week D3; Test type: Superiority or Other; p < .0001, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 5: Comparison: 2000 IU/Day D3 vs Vitamin D3 4000 IU/Day; Test type: Superiority or Other; p < .02, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 6: Comparison: 2000 IU/Day D3 vs 50,000 IU/Week D3; Test type: Superiority or Other; p < .0001, ANOVA; Bonferroni/Dunn adjustment
Statistical Analysis 7: Comparison: Vitamin D3 4000 IU/Day vs 50,000 IU/Week D3; Test type: Superiority or Other; p < .0003, ANOVA; Bonferroni/Dunn adjustment

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Vitamin D3 800 IU/Day | 2000 IU/Day D3 | Vitamin D3 4000 IU/Day | 50,000 IU/Week D3
Serious Adverse Events (participants affected / at risk) | 7/23 | 2/20 | 1/24 | 3/14
Other Adverse Events (participants affected / at risk) | 1/23 | 1/20 | 0/24 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 800 IU/Day (N=23) | 2000 IU/Day D3 (N=20) | Vitamin D3 4000 IU/Day (N=24) | 50,000 IU/Week D3 (N=14)
serious (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
flu/pneumonia/sepsis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
renal complication (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — biliary obstruction
fall + fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 800 IU/Day (N=23) | 2000 IU/Day D3 (N=20) | Vitamin D3 4000 IU/Day (N=24) | 50,000 IU/Week D3 (N=14)
ER visit (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
chest pain (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No